CLINICAL TRIAL: NCT03410966
Title: Paroxysmal Atrial Fibrillation Recurrences After Catheter Ablation: an Existing Correlation Between Oxidative Stress, Inflammation, Failing Heart Biomarkers and Atrial Fibrotic Remodeling.
Brief Title: Atrial Fibrillation Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Celestino Sardu, Clinical Professor, University of Campania Luigi Vanvitelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2712.2017
Record Dates: First submitted 2017-12-28; First posted 2018-01-25 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Atrial Fibrillation; Heart Failure, Diastolic
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure, Diastolic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): All patients affected by paroxysmal symptomatic atrial fibrillation, and anti-arrhythmic drug refractory atrial fibrillation will receive a trans catheter ablation therapy (intervention).
  Interventions: Procedure: trans cateheter ablation

INTERVENTIONS:
Procedure: trans cateheter ablation — All AF patients will receive trans catheter ablation by radiofrequency, to destroy arrhythmic atrial cells, and to isolate arrhythmic atrial firing around pulmonary veins' ostia.
  Other Names: magnetic resonance of left atrium

SUMMARY:
Objective. Atrial fibrillation (AF) recurrence after catheter ablation (CA) is a relevant clinical problem.

Methods. 123 patients with paroxysmal AF will be identified and screened for participation in this randomized, prospective, double blind, controlled placebo multicenter trial. 109 patients will be randomly assigned and enrolled in the study trial. Enrolled patients will receive magnetic atrial resonance and then will be treated by CA to receive pulmonary vein isolation (PVI). In this patients cytokines, inflammatory markers, and biomarkers such as ST2 protein and B type natriuretic peptide (BNP) will be evaluated at baseline, after CA, and during follow up. These biomarkers will be correlated to clinical outcomes (AF recurrences and heart failure progression and hospitalizations), and to fibrotic atrium extension as evaluated by magnetic resonance.

DETAILED DESCRIPTION:
Catheter ablation (CA) is first class treatment to restore sinus rhythm in patients with paroxysmal, symptomatic, drug refractory atrial fibrillation (AF). The sinus rhythm restoration after a successful CA may improve symptoms, New York Heart Association (NYHA) class and quality of life, reducing thromboembolic complications, and the likely progression of the arrhythmic disease towards forms of heart failure. Conversely, patients that do not respond successfully to CA therapy may still have AF, that is linked to an increased risk of ischemic stroke, heart failure, and overall mortality. AF recurrence after CA occurs in a percentage of patients ranging from 20% to 60%. This high rate of therapeutic failure, and the higher number of patients suffering for paroxysmal AF, represent a not acceptable problem in the clinical practice. The causes to explain this therapeutic failure are not completely clear, and broadly investigated by authors. To date, hyper activity of inflammatory tone, and oxidative stress with secondary left atrium enlargement and fibrosis, may represent a crucial part of molecular, and cellular adaptive processes linked to electro-anatomical remodeling, and to the AF perpetuation after an ablative treatment. Intriguingly, if the atrial fibrosis extension is a known process linked to worse prognosis, conversely the ablative approach therapy by burning to destroy arrhythmic cells, may also induce inflammation and atrial fibrotic lines around the veins' ostia. Therefore, the double face of the coin shows to the investigators the atrial fibrosis as an adaptive remodeling process linked to worse prognosis, and the atrial fibrosis as the result of a correct ablative approach to isolate pulmonary veins ostia and to improve clinical outcomes. To simply the concept, authors have to consider the first as an adaptive process leading to worse prognosis in AF patients, and the second as a necessary treatment to improve clinical outcomes in AF patients. Different studies have investigated cytokines, inflammatory markers, and other peptides such as B type natriuretic peptide (BNP), before and after CA in paroxysmal AF patients. These markers, and particularly BNP are correlated to atrial fibrosis extension, and worse prognosis after an ablative approach, and to the progression towards failing heart disease. Recently, the ST2 protein has been proposed as a new marker of heart fibrosis, such as a predictor of heart failure. Currently, no data has been reported about ST2 protein and AF recurrences after an ablative approach. Moreover, in the current study authors will investigate at baseline, and at follow up after an ablative approach, the using of cytokines, inflammatory markers, and other peptides such as B type natriuretic peptide (BNP), and ST2 protein, regards to these adaptive atrial fibrotic processes, and to AF recurrences after catheter ablation. Therefore, in this study authors will evaluate these biomarkers in patients with symptomatic and drug refractory paroxysmal AF undergoing catheter ablation interventions, and their correlation to AF recurrence rate after catheter ablation. To date, in the present study authors will correlate these biomarkers, and particularly ST2 protein to AF recurrences after CA, to left atrium fibrotic remodeling, and to hospitalizations events for heart failure at 12 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18,
* aged less than 75;
* clinical diagnosis of paroxysmal atrial fibrillation (AF)
* clinical diagnosis of symptomatic and anty- arrhythmic drugs refractory (AF)
* echocardiographic diagnosis of normal left atrium volumetry (left atrium volume < 30 ml/mq)
* echocardiographic diagnosis of normal left ventricle ejection fraction (LVEF) (LVEF > 55%).

Exclusion Criteria:

* aged less than 18,
* aged more than 75;
* clinical diagnosis of not paroxysmal AF;
* clinical diagnosis of heart failure;
* echocardiographic diagnosis of left atrium dilatation (left atrium volume > 30 ml/mq);
* echocardiographic diagnosis of LVEF depression (LVEF <55%).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Atrial Fibrillation (AF) recurrence | 12 months
  Authors will evaluate the percentage of patients in stable sinus rhythm after AF trans catheter ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Celestino Sardu, MD, MSc, PhD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Raffaele Marfella, Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 6 months